CLINICAL TRIAL: NCT00725504
Title: Effect of IV Lidocaine Infusions on Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sean Mackey, Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-07072008-1232
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain

ARMS (1):
- Lidocaine infusion (Experimental): Each participant will receive an intravenous infusion of lidocaine. Plasma concentrations will be increased gradually from 0-5 µg/ml.
  Interventions: Drug: Intravenous lidocaine

INTERVENTIONS:
Drug: Intravenous lidocaine — Intravenous lidocaine administered up to 5 µg/ml.

SUMMARY:
Our goals for this study involve using intravenous lidocaine as it is normally used in the Stanford Pain Management Center to assess the effect of intravenous lidocaine on chronic pain. Studies have been done determining the efficacy of intravenous lidocaine for treating pain but little research has been done to determine the effects of an intravenous lidocaine infusion on the different components of the pain experience. Our study will incorporate pain quality measures both before and during the infusions of lidocaine to determine changes in present pain intensity.

DETAILED DESCRIPTION:
Each patient will receive an intravenous infusion of lidocaine. Drug will be infused using a computer-controlled paradigm. This paradigm allows increasing plasma concentrations in a step-wise manner, keeping the concentration during each infusion step constant. Plasma concentrations will be increased gradually from 0 to 5 ug/ml in a method at the discretion of the medical team. This will be conducted according to standard medical practice for the infusion and the study procedures will not affect the infusion paradigm. Total infusion time is approximately 1-2 hours. During the course of the study, the primary outcome measure was changed from blood oxygenation level dependent (BOLD) signal to pain intensity.

ELIGIBILITY:
Inclusion Criteria:- subjects between the ages of 18 and 100 years for clinical component; subjects between the ages of 18 and 70 for the MRI component

* meets the study criteria of chronic pain of either peripheral or central origin
* male or a non-pregnant, non-lactating female. If females are of reproductive potential (i.e., not surgically sterilized and/or not post menopausal), they must be practicing an accepted method of birth control, agree to a urine pregnancy test at the start of each study session (for patient scheduled through the clinic, this has already been addressed by the recommending physician)
* is not currently on a sodium channel blocking agent, anticonvulsant, or tricyclic antidepressant,
* must be able to comply with any other study requirements and complete experimental tasks
* have no reported substance abuse within the past six months; Exclusion Criteria:- subject is lactating or pregnant;
* subject suffers from clinically significant cardiac, pulmonary, renal or liver disease;
* subject allergic to lidocaine.
* MRI Component: any metal objects (especially surgical clips), devices, or implants or any other MRI contraindication

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2008-09; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Mackey, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 71 patients were recruited through the Stanford University Pain Management Center.
Pre-assignment Details: Individuals were assessed for neuropathic pain prior to enrollment. Those with co-morbid cardiac disease were excluded from the study.
Groups:
- Lidocaine Infusion: Each participant will receive an intravenous infusion of lidocaine. Plasma concentrations will be increased gradually from 0-5 ug/ml.
  Intravenous lidocaine: Intravenous lidocaine administered during fMRI scan at a maximum dose of 3mcg/ml
Period: Overall Study
Arm/Group | Lidocaine Infusion
Started | 71
Completed | 71
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Seventy-one patients with chronic neuropathic pain
Arm/Group | Lidocaine Infusion
Number analyzed (Participants) | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 60
  >=65 years | 10
Age, Continuous [Mean (Full Range); unit: years] | 47 [17 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 39
Region of Enrollment [Number; unit: participants]
  United States | 71

OUTCOME MEASURES:

1. Primary Outcome: Present Pain Intensity
Description: Present pain intensity was measured using the visual analog scale (VAS). This is scored between 0 (no pain) to 10 (worst possible pain).
Time Frame: Patients completed the VAS of present pain intensity immediately before and immediately after placebo and during each infusion level
Measure: Mean (Standard Error); unit: Units on a scale
Groups:
- Baseline: Each participant was tested at the zero infusion rate.
- Placebo: Each participant received a placebo-saline infusion.
- Lidocaine 3 µg/ml: Each participant received an intravenous infusion of 3 µg/ml of lidocaine.
- Lidocaine 5 µg/ml: Each participant received an intravenous infusion of 5 µg/ml of lidocaine.
Arm/Group | Baseline | Placebo | Lidocaine 3 µg/ml | Lidocaine 5 µg/ml
Number analyzed (Participants) | 71 | 71 | 71 | 71
Units on a scale | 6.25 (0.23) | 5.64 (0.24) | 4.92 (0.27) | 4.18 (0.28)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the infusion period (approximately one hour) for each participant.
Description: The definitions for adverse event and serious adverse event did not differ from clinicaltrials.gov.
Arm/Group | Lidocaine Infusion
Serious Adverse Events (participants affected / at risk) | 0/71
Other Adverse Events (participants affected / at risk) | 9/71
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lidocaine Infusion (N=71)
Transient central nervous system side effects (General disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No